CLINICAL TRIAL: NCT03427632
Title: Role of Percutaneous Vertebroplasty in Treatment of Vertebral Tumors
Acronym: PVP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mustafa syd, Principal Investigator, Assiut University
Other Study IDs: PVPfortumors
Record Dates: First submitted 2018-01-29; First posted 2018-02-09 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Bone Tumor
Keywords: PVP; bone tumor
MeSH Terms: conditions — Bone Neoplasms | interventions — Bone Cements; Polymethyl Methacrylate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- percutaneous Vertebroplasty: patients meet the inclusion and exclusion criteria will be subjected to percutaneous vertebroplasty receiving bone cement (Polymethyl methacrylate)
  Interventions: Drug: Bone Cements

INTERVENTIONS:
Drug: Bone Cements — patents in PVP group will get injected with bone cement inside the collapsed malignant vertebra
  Other Names: Polymethyl methacrylate

SUMMARY:
Percutaneous vertebroplasty is a new technique to strengthen bone and reduce pain for patients with vertebral tumors

DETAILED DESCRIPTION:
Destructive vertebral lesions are a common in metastatic disease, multiple myeloma and lymphoma. Symptoms are caused by pathologic fracture consequences secondary to vertebral destruction, development of spinal instability and compression of adjacent neurological elements. Nonoperative treatments include radiotherapy, hormone therapy, cytotoxic drugs which are effective to halt the osteolytic process and reverse the neurological compromise, however; they cannot provide stability or relieve pain or cord compression. Surgical management options including vertebrectomy, reconstruction with a cage or PMMA bone cement, and stabilization with pedicle screws can restore spinal canal support and neurological functions also control pain, however; usually associated with high postoperative morbidity and mortality. Also not advisable for multifocal spinal disease. Percutaneous vertebroplasty is a new technique to strengthen bone and reduce pain. It is percutaneous, minimally invasive, image-guided procedure that involves injection of radio-opaque bone cement into a partially collapsed vertebral body, in an effort to provide stability and pain relief. The exact mechanism of pain relief remains unclear. Proposed theories include more favourable biomechanics after cement strengthening, chemical toxicity and exothermic effect of cement polymerization on nerve endings.

ELIGIBILITY:
Inclusion Criteria:

* Spinal instability
* Pain with movement
* Multiple level involvement
* Expected survival 3-6 months

Exclusion Criteria:

* Absolute
* Asymptomatic
* improving on medical treatment without worsening of the collapse.
* infection local or systemic
* uncorrectable coagulopathy
* Allergy to bone cement or contrast media
* Relative
* Radicular pain
* Tumor extension inside the vertebral canal or cord compression
* Fracture of the posterior column
* Sclerotic metastasis
* Diffuse metastases

Ages: 1 Year to 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Male or female patients diagnosed with vertebral body metastasis, multiple myloma, lymphoma meet the inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 11 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
pain relief | immediate
  reduction of spine pain following the injection of bone cement in the tumor according to Numeric Rating Scale, Improvement will be considered if NRS score decrease ≧ 20% after PVP

CONTACTS AND LOCATIONS:
Overall Officials: Nisreen Abbas, MD, Study Chair — Assiut University
Locations (1):
- Assiut University hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alvarez L, Perez-Higueras A, Quinones D, Calvo E, Rossi RE. Vertebroplasty in the treatment of vertebral tumors: postprocedural outcome and quality of life. Eur Spine J. 2003 Aug;12(4):356-60. doi: 10.1007/s00586-003-0525-z. Epub 2003 Mar 22. PMID 12687441
- [Background] Melton LJ 3rd, Kyle RA, Achenbach SJ, Oberg AL, Rajkumar SV. Fracture risk with multiple myeloma: a population-based study. J Bone Miner Res. 2005 Mar;20(3):487-93. doi: 10.1359/JBMR.041131. Epub 2004 Nov 29. PMID 15746994
- [Background] Wenger M, Markwalder TM. Re: Percutaneous vertebroplasty for pain relief and spinal stabilization (Spine 2000; 25: 923-8). Spine (Phila Pa 1976). 2000 Nov 15;25(22):2968-9. doi: 10.1097/00007632-200011150-00022. No abstract available. PMID 11074686
- [Background] Tsoumakidou G, Too CW, Koch G, Caudrelier J, Cazzato RL, Garnon J, Gangi A. CIRSE Guidelines on Percutaneous Vertebral Augmentation. Cardiovasc Intervent Radiol. 2017 Mar;40(3):331-342. doi: 10.1007/s00270-017-1574-8. Epub 2017 Jan 19. PMID 28105496